CLINICAL TRIAL: NCT07313085
Title: Physiopathogenic Mechanisms of Fecal Incontinence in Wolfram Syndrome
Brief Title: Mechanisms of Fecal Incontinence in Wolfram Syndrome
Status: Not yet recruiting | Type: Observational
Sponsor: Hôpital Necker-Enfants Malades (Other)
Responsible Party: Principal Investigator, Christophe Orssaud, Medical doctor, UF Ophthalmology HEGP
Other Study IDs: FECINCONTWS1125
Record Dates: First submitted 2025-11-15; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Wolfram Syndrome; Fecal Incontinence
MeSH Terms: conditions — Wolfram Syndrome; Fecal Incontinence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Wolfram syndrome patients with fecal incontience: wolfram syndrome patients without fecal incontinence
  Interventions: Other: Retrospective case-control analysis
- Wolfram syndrome patients without fecal incontience
  Interventions: Other: Retrospective case-control analysis

INTERVENTIONS:
Other: Retrospective case-control analysis — retrospective analysis of data

SUMMARY:
In order to clarify the mechanism of fecal incontinence in in Wolfram syndrome and to characterize its risk factors, the examiner will reviewed the files of patients followed in a Reference Center for Rare Diseases in Ophthalmology.

ELIGIBILITY:
Inclusion Criteria:

* Wolfram syndrome

Exclusion Criteria:

* no information concerning fecal incontinence in data records

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: retrospectif cohort of the rare disease center
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Urinary disorders | The date at the baseline
  number of patients with urinary disorder in each group according to the group

SECONDARY OUTCOMES:
sleep apnea | The date the data will be analyzed at the baseline
  number of patients with sleep apnea in each group according to the group
frequence of swallowing disroder | The data will be analyzed at baseline
  number of patients with swallowing disorders in each group according to the group
frequence of diabetes insipidus | The data will be analyzed at baseline
  number of patients with diabetes insipidus in each group according to the group
mutation type | The data will be analyzed at baseline
  report of mutations of WFS1 in each group

CONTACTS AND LOCATIONS:
Locations (1):
- HEGP, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided